CLINICAL TRIAL: NCT04331457
Title: Predictors Of Stroke Outcome In Children Admitted To Assiut University Children Hospital
Brief Title: Predictors Of Stroke Outcome In Chidren
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahlam Abdelbast Mohamad, principal investigator, Assiut University
Other Study IDs: posoicauch
Record Dates: First submitted 2019-09-24; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2019-09

CONDITIONS: Ischemic Stroke; Hemorrhagic Shock
Keywords: Seizures; Coma,; Altered mental status; Headache
MeSH Terms: conditions — Ischemic Stroke; Shock, Hemorrhagic; Seizures; Coma; Headache | interventions — Magnetic Resonance Spectroscopy; Blood Cell Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Brain magnetic resonance imaging (MRI) , computed tomography (CT) — imaging
  Other Names: complete blood count , echocardiography

SUMMARY:
Stroke can be defined as an abrupt loss of brain function that is caused by decreased cerebral blood flow.

Stroke can occur at all stages of life, but presentation is variable depending on age, involved artery, and underlying risk factors.

DETAILED DESCRIPTION:
Introduction Stroke can be defined as an abrupt loss of brain function that is caused by decreased cerebral blood flow.

Stroke can occur at all stages of life, but presentation is variable depending on age, involved artery, and underlying risk factors.

Younger children usually present with non specific symptoms such as seizures and altered mental status, especially those younger than 1 year, whereas older children present with focal neurologic deficits such as hemiplegia.(Rosa M et al ., 2016) Types pediatric stroke can be divided into ischemic and hemorrhagic stroke. Ischemic stroke is defined as focal damage to an area of brain tissue within a vascular territory due to loss of blood flow or oxygenation. It differs from diffuse hypoxic-ischemic injury in its mechanisms and distribution. Ischemic stroke, which represents 55% of pediatric strokes, can be subdivided into injuries caused by arterial ischemic stroke (AIS), which is due to loss of arterial flow, or venous infarction, which is due to loss of flow in a draining cerebral vein or venous sinus. Cerebral sinovenous thrombosis (CSVT), which involves obstruction by clot of a major venous sinus draining the brain parenchyma, can lead to infarcted brain parenchyma; Hemorrhagic stroke includes spontaneous hemorrhage within the brain parenchyma (intraparenchymal hemorrhage) and spontaneous (nontraumatic) subarachnoid hemorrhage. (Miya E et al.,2016) Risk factors Risk factors for stroke in children differ from those in adults. Adult risk factors are centered mainly on obstructive atherosclerotic, arteriopathies, cardiovascular disease, and arrhythmias, which are seldom found as risk factors in children. Stroke in children occurs primarily through 2 mechanisms, ischemic and hemorrhagic.

The most common cause of ischemic stroke is thrombotic, which occurs more commonly in children, representing 30% to 60% of cases. Although less common in children, hemorrhagic stroke is mainly caused by arteriovenous malformation.1 Studies such as the International Pediatric Stroke Study (IPSS) have reported systemic risk factors for pediatric stroke including sickle cell disease, cardiac disorders, trauma, and major infections such as meningitis, sepsis, and encephalitis, but in most cases, no systemic disease was found.(Rose M et al ., 2015) &(Simma B et al., 2013) Outcome of stroke Outcome of arterial ischemic stroke (AIS) in children is considered more favorable than in adults due to the better brain plasticity in children. However, several studies showed that more than half of survivors of childhood AIS have long-term physical disabilities and cognitive impairment. (Studer M et al .,2014) Although stroke etiolog and risk factors were different, stroke severity and clinical outcomes were similar (Bigi S et al .,2011) younger age at stroke is associated with poorer intellectual outcome and a broader spectrum of dysfunctions across multiple neuropsychological domains.(Allman C et al.,2013) Further, children with combined cortical and subcortical lesions have overall poorer cognitive outcome,(Westmacott R et al,.2010) larger lesion size negatively influences cognitive and functional outcome, possibly due to disruption of more neural network connections, adversely affecting functional brain organization.(Long B et al., 2011).

Regarding lesion laterality, controversial reports exist concerning the effect of lesion laterality on neuropsychological outcome. In addition, persistent seizures and persistent NI such as hemiplegia/paresis or visual field deficits also negatively influence neuropsychological and functional outcome. . (Allman C et al.,2013) NeuroImaging Brain magnetic resonance imaging (MRI) as more sensitive than computed tomography (CT) in diagnosis and detection of pediatric stroke. Head CT without contrast is the study of choice for identifying acute hemorrhage but may be normal in the cases of ischemic stroke in the first 12 to 24 hours after the event .( Alberts MJ et al., 2011)& (Elbers J et al.,2015) Therefore, MRI is a more sensitive modality for stroke including AIS, vascular malformations, and central nervous system inflammatory changes. Non contrast CT used for the detection of brain ischemia is more sensitive after the initial 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* - Infant and Children around age of (1month to 18years old) of both sexes were diagnosed as stroke (hemorrhagic or ischemic) by CT or MRI.

Exclusion Criteria:

* - Neonates (less than one month)
* Stroke caused by trauma
* Patient refusal to participate the research

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: infant and children diagnosed as stroke by CT brain and MRI brain
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Computed tomography(CT) of the brain | Baseline to 6 months after discharge
  To detect the stroke type ;(hemorrhagic or ischemic) , location and severity at admission (at start of the study) and after discharge (6 months after discharge) .
Brain magnetic resonance imaging (MRI) | 1Year
  It is more sensitive than brain CT in diagnosis and detection of pediatric stroke including AIS , vascular malformations , and central nervous system inflammatory changes.
Glasgow coma scale(GCS). | 1 year
  To assess the level of consciousness to evaluate the extent of brain damage;(15_12) mild brain damage,(12_8) moderate brain damage,(<8 )severe brain damage.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goeggel Simonetti B, Cavelti A, Arnold M, Bigi S, Regenyi M, Mattle HP, Gralla J, Fluss J, Weber P, Hackenberg A, Steinlin M, Fischer U. Long-term outcome after arterial ischemic stroke in children and young adults. Neurology. 2015 May 12;84(19):1941-7. doi: 10.1212/WNL.0000000000001555. Epub 2015 Apr 10. PMID 25862797
- [Background] Studer M, Boltshauser E, Capone Mori A, Datta A, Fluss J, Mercati D, Hackenberg A, Keller E, Maier O, Marcoz JP, Ramelli GP, Poloni C, Schmid R, Schmitt-Mechelke T, Wehrli E, Heinks T, Steinlin M. Factors affecting cognitive outcome in early pediatric stroke. Neurology. 2014 Mar 4;82(9):784-92. doi: 10.1212/WNL.0000000000000162. Epub 2014 Jan 31. PMID 24489131
- [Background] McKinney SM, Magruder JT, Abramo TJ. An Update on Pediatric Stroke Protocol. Pediatr Emerg Care. 2018 Nov;34(11):810-815. doi: 10.1097/PEC.0000000000001653. PMID 30395072
- [Background] Chiang KL, Cheng CY. Epidemiology, risk factors and characteristics of pediatric stroke: a nationwide population-based study. QJM. 2018 Jul 1;111(7):445-454. doi: 10.1093/qjmed/hcy066. PMID 29648667